CLINICAL TRIAL: NCT00939393
Title: ESS Performed in Operating Room Versus Clinician's Office
Brief Title: Balloon Sinus Dilation In Office or OR
Acronym: ORIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPR005002
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- FESS in OR with or without balloons (Active Comparator): Functional Endoscopy Sinus Surgery
  Interventions: Device: FESS instruments with or without balloon treatment
- Balloon sinuplasty in physician office (Active Comparator): Balloon Sinuplasty in physician office using Acclarent devices
  Interventions: Device: Balloon Sinuplasty

INTERVENTIONS:
Device: FESS instruments with or without balloon treatment — Intervention with metal instruments with or without balloon treatment
  Arms: FESS in OR with or without balloons
Device: Balloon Sinuplasty — Balloon dilatation of sinuses
  Arms: Balloon sinuplasty in physician office

SUMMARY:
Endoscopic sinus surgery will be performed either in the physician's office or in the operating room (OR). Patients treated in the physician's office will have endoscopic sinus surgery performed with balloon sinuplasty devices. Patients treated in the OR will have endoscopic sinus surgery performed with or without balloon sinuplasty devices.

DETAILED DESCRIPTION:
In this study, endoscopic sinus surgery will be performed either in the physician's office or in the operating room (OR). Patients treated in the physician's office will have endoscopic sinus surgery performed with the balloon sinuplasty devices. Patients treated in the OR will have endoscopic sinus surgery performed with or without balloon sinuplasty devices. Both primary treatment of sinusitis as well as revision of previously treated sinuses will be allowed. Resource absorption will be evaluated for both venues.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and greater
2. Both male and female patients eligible
3. Diagnosis of chronic sinusitis that is not responsive to medical management (> 12 weeks of symptoms and failed at least 3 to 6 weeks of appropriate antibiotic therapy as evidenced by presence of disease on CT scan)
4. Planned endoscopic sinus surgery (recommended by investigator, consented to by patient)

Exclusion Criteria:

1. Cystic fibrosis
2. Samter's Triad (Aspirin sensitivity, Asthma, Sinonasal polyposis)
3. Sinonasal tumors or obstructive lesions
4. History of facial trauma that distorts sinus anatomy and precludes access to the sinus ostium
5. Ciliary dysfunction
6. Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levine, MD, Principal Investigator — Rockside Road Surgery Center Independence, OH
Locations (1):
- Rockside Road Surgery Center, Independence, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients presenting to the study sites (medical clinics) for whom endoscopic sinus surgery was recommended were offered the opportunity to participate in the study by study investigators.
Groups:
- In Office: Endoscopic sinus surgery performed in physician's office using balloon sinus dilation device.
- Operating Room: Endoscopic sinus surgery performed in the operating room (OR) with or without balloon sinus dilation devices.
Period: Overall Study
Arm/Group | In Office | Operating Room
Started | 37 | 35
Completed | 33 | 35
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Office: Endoscopic sinus surgery performed in physician's office using balloon sinus dilation device.
- Total: Total of all reporting groups
Arm/Group | Office | Operating Room | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.5) | 47.5 (15.1) | 51.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 37 | 35 | 72

OUTCOME MEASURES:

1. Secondary Outcome: Mean Intra-patient Change in Lund-MacKay CT Score [24 Weeks]
Description: The Lund-MacKay (LMK) CT (computed tomography) score is a scoring system to evaluate radiographic opacification of the paranasal sinuses. The LMK score will be evaluated at 24 weeks post-procedure compared to baseline. The LMK scoring system rates each of both the left and right frontal, maxillary, sphenoid, ostiomeatal complex, anterior ethmoid and posterior ethmoid sinuses on a scale of 0 to 2, where '0' is 'no opacification' and '2' is 'complete opacification'. The scores for a given subject are totaled and expressed as the LMK score, where zero is the minimum score, and 24 is the maximum score. A higher score represents greater sinus disease burden.
Time Frame: 24 weeks
Population: Eight (8) In-Office subjects and 15 Operating Room subjects were missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 29 | 20
Scores on a scale | -3.83 (4.08) | -5.65 (5.27)

2. Secondary Outcome: Proportion of Participants Rating Procedure as Tolerable (IO Only)
Description: Participants evaluated the tolerability of their balloon dilation in office (IO = In Office) procedure on a scale from zero to 5, where '0' represented 'not tolerated' and '5' represented 'highly tolerable'. Scores of 3 through 5 were consdered tolerable ratings. The endpoint reports the proportion of participants rating the procedure as tolerable.
Time Frame: Day 0
Population: Eight (8) In-Office subjects were missing data for this outcome measure.
Measure: Number; unit: participants
Arm/Group | In Office
Number analyzed (Participants) | 29
participants | 27

3. Secondary Outcome: Proportion of Participants Reporting No Pain or Pain of Low Intensity (IO Only)
Description: Participants evaluated the per-procedural pain of their balloon dilation in office (IO = In Office) procedure on a scale from zero to 5, where '0' represented 'no pain' and '5' represented 'intense pain'. Scores of 0 through 2 were considered ratings of no pain or pain of low intensity. The endpoint reports the proportion of participants reporting no pain or pain of low intensity.
Time Frame: Day 0
Population: One (1) In-Office subject was missing data for this outcome measure.
Measure: Number; unit: participants
Arm/Group | In Office
Number analyzed (Participants) | 36
participants | 24

4. Secondary Outcome: Mean Number of Debridements Per Participant (IO Only)
Description: A debridement is a procedure to remove post-surgical crusts, mucus, and fibrin from obstructed nasal and sinus cavities after functional endoscopic sinus surgery. Each physician visit in which a debridement was performed was counted as one debridement.
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: debridements
Arm/Group | In Office
Number analyzed (Participants) | 37
debridements | 0.42 (0.51)

5. Secondary Outcome: Proportion of Participants With Revisions (IO Only)
Description: After sinus surgery, the patient may require a subsequent sinus procedure (a revision procedure) to address recurrence of disease. These revision procedures are assessed in this outcome measure.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | In Office
Number analyzed (Participants) | 37
participants | 1

6. Secondary Outcome: Proportion of Participants With Post-operative Sinus Infections
Description: Investigators reported the sinus infections as secondary to chronic rhinosinusitis (CRS) or other pre-existing conditions such as allergies. The rates of these sinus infections are consistent with the disease burden of the subjects and consistent with post procedure symptomatology associated with endoscopic sinus surgery (ESS).
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 37 | 35
participants | 13 | 12

7. Secondary Outcome: Mean Intra-patient Change in SNOT-20 Score at 1 Week Post-procedure Compared to Baseline
Description: The 20 question Sino-Nasal Outcome Test (SNOT-20) will be used to evaluate sinus symptoms and sinus-symptom related quality of life (QOL) at baseline, 1 week, 4 weeks, 24 weeks and 52 weeks post-procedure. The change in SNOT-20 score at each post-procedure time point will be evaluated compared to baseline SNOT-20 score. Each of the 20 questions in the SNOT-20 survey is scored on a scale of 0 to 5, where '0' represents 'no problem' and '5' represents 'problem as bad as it can be'. The 20 questions are expressed as a mean of the scores. Therefore, the minimum mean score is zero and the maximum mean score is 5.
Time Frame: 1 week
Population: Five (5) In-Office subjects and 2 Operating Room subjects were missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 32 | 33
scores on a scale | -0.98 (0.79) | -0.71 (1.07)

8. Secondary Outcome: Mean Intra-patient Change in SNOT-20 Score at 4 Weeks Post-procedure Compared to Baseline
Description: as for outcome 7
Time Frame: 4 weeks
Population: Six (6) In-Office subjects and 2 Operating Room subjects were missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 31 | 33
scores on a scale | -1.32 (0.89) | -1.21 (1.12)

9. Secondary Outcome: Mean Intra-patient Change in SNOT-20 Score at 52 Weeks Post-procedure Compared to Baseline
Description: as for outcome 7
Time Frame: 52 weeks
Population: Sixteen (16) In-Office subjects and 24 Operating Room subjects were missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 21 | 11
scores on a scale | -1.43 (0.96) | -1.10 (1.05)

10. Primary Outcome: Mean Intra-patient Change in SNOT-20 Score at 24 Weeks Post-procedure Compared to Baseline
Description: as for outcome 7
Time Frame: 24 weeks
Population: Eleven (11) In-Office subjects and 10 Operating Room subjects were missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- In Office: Endoscopic sinus surgery (ESS) performed in physician's office (IO, or In Office) using balloon sinus dilation device.
- Operating Room: Endoscopic sinus surgery (ESS) performed in the operating room (OR) with or without balloon sinus dilation devices.
Arm/Group | In Office | Operating Room
Number analyzed (Participants) | 26 | 25
scores on a scale | -1.25 (0.99) | -1.35 (1.12)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.
Arm/Group | Office | Operating Room
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 1/37 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Office (N=37) | Operating Room (N=35)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.
Swallowed pledget (Gastrointestinal disorders) | 1 (1) | 0 (0) — Adverse event assessment by physician according to defined follow-up visit schedule, and by patient self-reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days